CLINICAL TRIAL: NCT02172976
Title: Randomized Multicenter Phase II/III Study With Adjuvant Gemcitabine Versus Neoadjuvant/Adjuvant FOLFIRINOX in Resectable Pancreatic Cancer
Brief Title: Randomized Multicenter Phase II/III Study With Adjuvant Gemcitabine Versus Neoadjuvant / Adjuvant FOLFIRINOX for Resectable Pancreas Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEPAFOX
Record Dates: First submitted 2014-05-23; First posted 2014-06-24 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Resectable Prancreas Carcinoma
Keywords: pancreas cancer; neoadjuvant chemotherapy; Folfirinox; gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin; Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFIRINOX (Experimental): Oxaliplatin 85mg/m², Irinotecan 180mg/m², 5-FU 400mg/m² Bolus i.v., 5-FU continuous Infusion 2400 mg/m² Natriumfolinate 400mg/m² 46h d1; qd15 6 cycles pre- and 6 cycles post- surgery
  Interventions: Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Irinotecan; Drug: Natriumfolinate
- Gemcitabine (Active Comparator): Gemcitabine 1000 mg/m² d1, d8, d15; qd 29; 6 cycles after surgery
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine
  Arms: Gemcitabine
Drug: Oxaliplatin
  Arms: FOLFIRINOX
Drug: 5-Fluorouracil
  Arms: FOLFIRINOX
Drug: Irinotecan
  Arms: FOLFIRINOX
Drug: Natriumfolinate
  Arms: FOLFIRINOX

SUMMARY:
In this multicenter study, patients with resectable pancreatic carcinoma will be treated with (a) surgery followed by 6 cycles gemcitabine or (b) 4-6 cycles FOLFIRINOX followed by surgery followed by 4-6 cycles FOLFIRINOX.

The overall survival between both therapies will be compared as well as other parameters.

DETAILED DESCRIPTION:
This is a phase II/III randomized multicenter study. Patients with resectable pancreatic carcinoma will be randomized in Arm A (surgery plus adjuvant gemcitabine, 6 cycles) or Arm B (4-6 cycles FOLFIRINOX neoadjuvant, 4-6 cycles FOLFIRINOX adjuvant).

Primary endpoint is the overall survival, secondary endpoints are progression-free survival, perioperative morbidity and mortality, rate of R0 resections, tolerability and feasibility of neoadjuvant FOLFIRINOX and others.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the pankreas. For histological confirmation, max. 3 tests are allowed. If no confirmation of carcinoma is possible, the patient can not be included into the study.
2. Radiological confirmation of a locally limited curativ resectable (primarily resectale or borderline situation) pankreas carcinoma without distant metastases.
3. no prior pancreas resection
4. no prior cytostatic chemotherapy
5. female and male patients > 18 and <=75 years using contraception
6. ECOG ≤ 1
7. medical resectability
8. granulocytes > 1.500/µl
9. thrombocytes > 100.000/µl
10. hemoglobin ≥ 8,0 g/dl
11. serumcreatinine ≤ 1.5x of normal value or Creatinine-Clearance > 50 ml/min
12. written informed consent

Exclusion Criteria:

1. Endocrine pancreas carcinoma
2. locally advanced inoperable stages: non-resectable infiltration of V. porta or longway infiltration of A. mesenterica superior or infiltration of Truncus coeliacus.
3. distant metastases
4. Relapse
5. prior radiotherapy of measurable lesions
6. peritonealcarcinosis
7. malignant secondary disease, dated back < 5 years (exeption: in-situ-carcinoma of the cervix, adequately treated skin basal cell carcinoma)
8. contraindication for operative resection
9. ECOG ≥ 2
10. severe liver dysfunction (AST/ALT>3,5xULN, AP>6xULN)
11. Transhepatic drainage
12. active CHD (symptoms present), cardiomyopathy or heart insufficiency stage III-IV according to NYHA and EF < 45%
13. severe non-surgical accompanying diseases or acute infection
14. chronic diarrhea
15. chronic inflammable gastro-intestinal disease
16. peripheral polyneuropathy > NCI grade II
17. pregnancy or lactation
18. hypersensibility or contraindication for Gemcitabine, Oxaliplatin, Natriumfolinate, Irinotecan or 5-Fluorouracil
19. participation in another interventional trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2020-01 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
median overall survival | From date of randomization until the date of death from any cause assessed up to 24 months

SECONDARY OUTCOMES:
median progression-free survival (PFS) | From date of randomization until the date of first documented progression / relapse or date of death from any cause, whichever came first, assessed up to 24 months
perioperative morbidity and mortality | 30 days after surgery
R0 resection rate | 2 months after surgery
pathological complete remission | at surgery
  during surgery, paraffin embedded tissue is prepared for analysis which is analyzed for remission grading at the central pathology afterwards
adverse events (grade, number per patient) related to of G-CSF prophylaxis in the Folfirinox arm | up to 40 weeks
prevalence of iron deficiency | baseline, d1 of every cycle, end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof., Principal Investigator — Institute of Clinical Cancer Research (IKF), UCT - University Cancer Center, Frankfurt, Germany
Locations (1):
- Institute of Clinical Cancer Research (IKF), UCT - University Cancer Center, Frankfurt, Germany, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- See also: Related Info — http://www.ikf-nordwest.de/